CLINICAL TRIAL: NCT03982602
Title: Safety and Feasibility of Ketogenic Diet for Traumatic Brain Injury Study Protocol
Brief Title: Ketogenic Diet for Traumatic Brain Injury
Acronym: KETI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Niraj Arora, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014675
Record Dates: First submitted 2019-06-03; First posted 2019-06-11 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury; Ketogenic Dieting
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects on Ketogenic diet (Experimental): Treatment with KD will consist of 4:1 [fat]: [protein + carbohydrate] weight ratio. KD will be started as soon as the patient is ready for alimentation (while they are in neurocritical care unit). The rate of feeds will be calculated by trained dietician on service. Ketogenic diet will be continued during the entire length of ICU stay. Supplementation with vitamins, calcium and phosphorus will be done.
  Interventions: Other: Ketogenic diet

INTERVENTIONS:
Other: Ketogenic diet — Subjects will be provided with the Ketogenic diet in the form of tube feeds once the decision is made to start the patient on diet.
  Other Names: Ketovie

SUMMARY:
Traumatic Brain Injury is a major health concern in United States. There is a un-met need to develop new therapeutic options for faster neuron recovery without causing significant side effects. The role of ketones in neuronal recovery has been studied and has been found to be useful in decreasing size of contusion. The present study aims to study the safety and feasibility profile of ketogenic diet.

DETAILED DESCRIPTION:
Traumatic Brain Injury (TBI) is a major health concern for United States contributing nearly one-third of injury-related deaths in United States. The Centers for Disease Control and Prevention (CDC) estimates that 1.7 million people in the United States sustain a TBI each year. It is responsible for significant disabilities and the total cost of productivity loss was estimated to be $76.5 billion in the United States in 2004.

Several animal models have demonstrated the effectiveness of ketones in brain injury to decrease the size of contusion, improving cortical ATP levels, reduced brain edema and cellular apoptosis. Ketones have been shown to be effective in neuromodulation in animal models. Evaluation of carbohydrate free diet has been done in traumatic brain injury patients and it was noted to not cause fluctuations in blood glucose. There is a need for safety and feasibility study of ketogenic diet in traumatic brain injury patients and to understand the effectiveness in neuromodulation in humans. The present study focuses on identifying the safety and feasibility of KD in traumatic brain injury patients.

This pilot project data will be utilized to design future randomized clinical trials. Based on the safety data, further trials will be conducted to evaluate the effectiveness of KD in traumatic brain injury patients and its effectiveness in controlling elevated intracranial pressure. It will open the avenue for consideration of new treatment option for intracranial pressure management and functional recovery. From a nutrition perspective, Ketogenic diet might become the standard of care for this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Severe Traumatic Brain Injury
2. GCS<= 8 with severe head injury
3. Age more than 18years

Exclusion Criteria:

1. Diabetic Ketoacidosis
2. Unstable metabolic condition (persistent hyponatremia, hypernatremia, hypoglycemia, hypocalcemia, acidosis)
3. Cardiorespiratory or hemodynamic instability
4. Coagulopathy
5. Pancreatitis
6. Liver Failure
7. Severe hyperlipidemia
8. Inability to tolerate enteral feeds including ileus
9. Known Fatty acid oxidation disorder or pyruvate carboxylase deficiency
10. Any terminally ill patient with poor brain stem reflexes and mortality within 24h of admission.
11. Pregnant Females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Effect of Ketogenic Diet on Intracranial Pressure | Baseline, till patient on KD (maximim 1 month)
  Intracranial Pressure will be measured hourly and it will be trended daily.
Development of Ketosis in blood | Baseline, till patient on KD ( maximum 1month)
  Serum beta-hydroxybutyrate will be done alternate day to assess the level of ketosis in blood.
Excretion of Ketones in Urine | Baseline, till patient on KD (maximum 1 month)
  Urine Ketones will be measured alternate day to assess the level of ketosis

SECONDARY OUTCOMES:
Evaluate change in the neurological exam | Baseline, before discharge from ICU
  Neurological exam will be documented with Glasgow Coma Scale.
Evaluate subjects with gastro-intestinal adverse effects | Baseline, till patient on KD (Maximum 1month)
  Adverse effects like Diarrhea, vomiting, abdominal distension (ileus), abdominal tenderness will be monitored.
Evaluate subjects for muscle wasting | Baseline, till patient on Kd (Maximum 1month)
  Urinary Nitrogen and urinary creatinine will be measured alternate day to look for muscle wasting.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arora N, Litofsky NS, Golzy M, Aneja R, Staudenmyer D, Qualls K, Patil S. Phase I single center trial of ketogenic diet for adults with traumatic brain injury. Clin Nutr ESPEN. 2022 Feb;47:339-345. doi: 10.1016/j.clnesp.2021.11.015. Epub 2021 Nov 16. PMID 35063224